CLINICAL TRIAL: NCT04201756
Title: Neoadjuvant Afatinib Therapy for Potentially Resectable Stage III EGFR Mutation-Positive Lung Adenocarcinoma: A Single-Arm, Open-Label, Phase II Clinical Trial
Brief Title: Neoadjuvant Afatinib Therapy for Potentially Resectable Stage III EGFR Mutation-Positive Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of science and education department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.0328(TEAM, LungMate-004)
Record Dates: First submitted 2019-12-04; First posted 2019-12-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Lung Adenocarcinoma Stage III; EGFR Gene Mutation
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afatinib (Experimental)
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — ①Neoadjuvant treatment stage: the enrolled patients take afatinib at a dosage of 40mg per day, 8-16 weeks in total; and receive CT scan re-examination in the 4th/8th/12th post-therapy week.
  ②Surgical treatment stage: the patients who respond to alfatinib treatment (CR+PR) and the patients who do not respond to alfatinib therapy but could still undergo surgery (SD and PD) will receive radical lung lobectomy+systematic lymph node dissection.
  ③Adjuvant treatment stage: The CR, PR and SD patients who have been treated surgically will take alfatinib at a dosage of 40mg per day for at least 1 year. The SD and PD patients who could not receive operation and the PD patients who have received operation will be transferred into medical oncology or/and radiation oncology and receive comprehensive therapy (chemotherapy or/and radiotherapy, the regimen is designed by oncologist and radiologist)

SUMMARY:
In general, for patients with stage I or II disease, surgery provides the best chance for cure.EGFR tyrosine kinase inhibitors(TKIs)are standard first-line treatment for EGFR-mutant advanced NSCLC.Afatinib was a 2nd-generation EGFR TKI that covalently bound and irreversibly blocked signaling through activated EGFR, human epidermal growth factor receptor 2 (HER2), and ErbB4 receptors, and the FDA has approved afatinib for first-line treatment of patients with metastatic NSCLC who have sensitizing EGFR mutations.The treatment of stage III NSCLC remains a matter of debate. Current multimodality treatment options for stage III included definitive chemoradiation, surgery followed by adjuvant therapy,or neoadjuvant therapy followed by surgical resection.Previous studies have revealed that adjuvant EGFR-TKI could significantly prolong disease free surivival, and have less toxicity than adjuvant chemotherapy for early resectable EGFR mutation positive NSCLC patients.EMERGING-CTONG1103 regarding neoadjuvant erlotinib vs chemotherapy (Gemcitabine plus cisplatin) for stage III NSCLC reveal that erlotinib has improved ORR (54%), major pathological response, operation rate, R0 resection and lymph node downstaging, and progression-free survival (PFS).A phase II trial (ASCENT) of neoadjuvant afatinib for stage III EGFR-mutation NSCLC concludes that afatinib yields the highest ORR (75%) up to now and verifies the feasibility of neoadjuvant EGFR TKIs for stage III NSCLC. However, no more studies are available so far to confirm the efficacy and safety of neoadjuvant afatinib in the treatment of resectable stage III EGFR mutation-positive NSCLC, and there is a lack of studies based on the Chinese population. Given that the neoadjuvant therapy has delayed the operation time and there is a potential risk of cancer progression, more data are needed to perform evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Lung adenocarcinoma patient with EGFR sensitive mutation as confirmed by needle biopsy;
* At stage III (TNM Staging, Version 8) as identified by chest CT, PET-CT or/and EBUS;
* No systemic metastasis (confirmed by head MRI, whole body bone scan, PET-CT, liver and adrenal CT, etc.);
* With the feasiblility or potential feasibility to receive radical surgery (radical lung lobectomy+systematic lymph node dissection);
* Good lung function that could tolerate surgical treatment;
* Aged >= 18 years;
* At least one measurable tumor foci (the longest diameter measured by CT shall be > 10 mm);
* Other major organs shall function well (liver, kidney, blood system, etc.):
* ECOG PS score shall be 0-1;
* The child-bearing female must undergo pregnancy test within 7 days before starting the treatment and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 30 days after completion of the trial. The child-bearing male shall use condom for contraception during the trial and within 30 days after completion of the trial;
* The patient shall sign the Informed Consent Form.

Exclusion Criteria:

* The patient has undergone any systemic anti-cancer treatment for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment, etc.;
* The patient suffered from other cancers besides NSCLC (except cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor [including Ta and Tis]) within 5 years before the trial;
* The patient suffers from any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina pectoris, angina pectoris that starts to attack within the last 3 months, congestive heart failure [≥ Grade II specified by New York Heart Association (NYHA)], cardiac infarction (6 months before enrollment), severe arrhythmia and liver, kidney or metabolic diseases that requires drug treatment;
* The patient is a carrier of active hepatitis B, hepatitis C or HIV;
* The patient suffers from severe or new-onset gastrointestinal diseases with diarrhea as the main symptom;
* The patient is receiving the P glycoprotein inhibitor therapy;
* The patient has had or is currently suffering from cardiovascular malformation;
* The patient has had or is currently suffering from interstitial lung disease;
* The patient had undergone other major systemic operations or suffered from severe trauma within 3 months before the trial;
* The patient is allergic to afatinib or its any excipients;
* The patient suffers from nervous system diseases or mental diseases and cannot keep compliance with the trial;
* The patient has any malabsorption condition;
* The female patient is in pregnancy or lactation period;
* There are any conditions under which the investigator considers the patient is not suitable to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 11 weeks
  ORR is defined as the proportion of patients who have completed the 8- to 16-week treatment with afatinib before operation and have achieved CR or PR as confirmed by CT evaluation after 3 weeks in all patients.

SECONDARY OUTCOMES:
Event-free survival (EFS) | up to 60 months
  It is was defined as the time from the first administration of afatinib in this study to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause (including any cause of death in the event of no progression)
Disease free survival (DFS) | up to 100 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression.
Overall survival (OS) | up to 60 months
  It is defined as the time from random enrollment to death of participant due to any cause.
Progression-free survival (PFS) | up to 60 months
  It is defined as the time from the first administration of afatinib in this study to the disease progression or death.
R0 resection | 9 weeks
  It is defined as the proportion of patients with negative surgical margin and no residual found under microscope after resection in all patients who have completed the treatment.
Pathological downstaging rate | 11 weeks
  It is defined as the proportion of patients who have completed the 8-week treatment with afatinib before operation and have achieved a T stage downing of the tumor as confirmed by CT evaluation after 3 weeks in all patients who have completed the treatment.
Treatment-related adverse events | 12 weeks
  It refers to the number of adverse events related to afatinib monotherapy or platinum-based chemotherapy as evaluated according to CTCAE v4.0.
Health related quality of life (HRQol) | 12 weeks
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shang'ai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.

REFERENCES:
- [Derived] Bian D, Sun L, Hu J, Duan L, Xia H, Zhu X, Sun F, Zhang L, Yu H, Xiong Y, Huang Z, Zhao D, Song N, Yang J, Bao X, Wu W, Huang J, He W, Zhu Y, Jiang G, Zhang P. Neoadjuvant Afatinib for stage III EGFR-mutant non-small cell lung cancer: a phase II study. Nat Commun. 2023 Aug 3;14(1):4655. doi: 10.1038/s41467-023-40349-z. PMID 37537219